CLINICAL TRIAL: NCT04776798
Title: The Effects of Biomechanical Taping on Individuals With Mechanical Low Back Pain With Increased Foot Pronation
Brief Title: Biomechanical Taping on Low Back Pain With Increased Foot Pronation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayse Zengin Alpozgen, Asst.Prof., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 05.SKHEK
Record Dates: First submitted 2021-02-27; First posted 2021-03-02 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Low Back Pain; Foot Posture; Taping; Functional Mitral Regurgitation
Keywords: biomechanical-taping; mechanical low back pain; foot posture; function
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biomechanical Taping (Experimental): Anti pronation taping will apply bilaterally with Dynamic Tape®. The tape will attach to the dorsal aspect of the foot.
  A home-based exercise program will apply in the first session. Printouts showing the exercises will give to the patients. Exercises will be done at home for 4 weeks, 5 d/w.
  Interventions: Other: Taping
- Placebo Taping (Placebo Comparator): Placebo Taping will apply bilaterally to each individual in the control group by the same physiotherapist, without any effect on increased pronation.
  A home-based exercise program will apply in the first session. Printouts showing the exercises will give to the patients. Exercises will be done at home for 4 weeks, 5 d/w.
  Interventions: Other: Taping

INTERVENTIONS:
Other: Taping — Tape applications will repeat twice per week, for 4 weeks.

SUMMARY:
It is stated that abnormal lower extremity posture and biomechanics are effective in the development and progression of Low Back Pain (LBP). Exercise, electrotherapy, insoles, and orthoses are used for the prevention and treatment of low back pain.The use of orthosis, insoles, and taping techniques stands out in the correction of foot posture and dysfunctions, which are stated to cause LBP. In studies examining the application of taping to improve foot posture and biomechanics, it is stated that taping is effective in improving foot posture and biomechanics in the short term.

Biomechanical taping has been used in the treatment of musculoskeletal disorders in recent years. It is aimed to correct the impaired joint biomechanics by reducing the load on the joint, supporting strength, and providing movement modification.

DETAILED DESCRIPTION:
In this study, it is assumed that correction of "increased foot pronation" with dynamic taping will result in the recovery of increased internal rotation and decreased shock absorption during weight-bearing, which is stated to cause pain. The study aims to investigate the effects of biomechanical tapping in combination with a home exercise program on LBP.

Participants with a diagnosis of LBP and bilateral increased flexible foot pronation will divide into two groups (Biomechanical Taping (BT) group or Placebo Taping (PT) group). Tape applications will repeat twice per week, for 4 weeks. And also a home-based exercise program will apply to both groups.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical low back pain for at least 6 months
* Age between 18-65 years
* Increased, bilateral, flexible pronation of the feet (Foot Posture Index-6 score> 0)

Exclusion Criteria:

* Rigid pes planus, pes cavus, equinus deformity, hallux valgus, hallux rigid or calcaneal epin in the feet
* Lower extremity injury or surgery in the last 6 months
* Radicular type back pain (patients with leg pain> low back pain)
* Body Mass Index (BMI)> 30,
* Use of analgesics
* Pregnancy
* Presence of symptoms related to a history of spinal surgery in the last 5 years.
* Neurological impairment or cognitive dysfunction (stroke, dementia, etc.)
* Rheumatological diseases
* Peripheral vascular diseases
* Difference in length between extremities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 4 week
  It is used to evaluate the level of pain.The activity, rest and night pain levels of the patients will be question.
Foot Posture Index (FPI-6) | 4 week
  FPI-6 examines foot posture under 6 headings: talar head palpation, supra and infra lateral malleoli curvature, calcaneal frontal plane position, prominence in region of talonavicular joint, congruence of medial longitudinal arch, abduction/adduction of forefoot on rearfoot. Each measure is scored from -2 to 2. A total score of 0 is considered a neutral foot; a positive score is for pronated foot, whereas a supinated foot is given a negative score.

SECONDARY OUTCOMES:
6 Minute Walk Test (6MWT) | 4 week
  The 6MWT provides an indirect assessment of physical performance and endurance capacity.the person is asked to walk for 6 minutes as fast as possible in the 30-meter straight corridor, the patient does not speak during walking, but is supported with motivating sentences at the end of every 1 minute. After 6 minutes, the distance traveled (meters-m) is recorded.
Step-On-Stool Test | 4 week
  The person tested is asked to step up onto and down from a stool at a self-selected speed. The step height is 0.40 meters for women, 0.44 meters for men. The number of steps managed will be record.
PILE Lumbar Lifting Test | 4 week
  The lumbar Spine is tested by asking to lift the box with a weight of 76 cm shelf from the ground to waist level. The test starts with weights of 3.6 kg for women and 5.9 kg for men. It is asked to lift the box containing weight 4 times in 20 seconds. For each completed round, a weight of 2.25 kg for women and 4.5 kg for men are added to the box. If the patient reaches 85% of the maximum heart rate, lifts 55-60% of his body weight, shows pain or fatigue after a 20-second interval, and cannot complete 4 repetitions within 20 seconds, the test is terminated. The maximum weight lifted & the number of repetitions multiplied so total work done will calculate and record.
Revised Oswestry Disability Index | 4 week
  ; It is a self-administered questionnaire and consists of 10 sections. Each section is scored between 1 and 5 (the highest score for the last question is 6), test scores range from 0 to 51. An increase in the score is interpreted as an increase in disability

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Zengin Alpozgen, PhD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Ayşe Alpözgen, Küçükçekmece, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No